CLINICAL TRIAL: NCT05843708
Title: A Phase 1, Open-Label Study to Evaluate the Effect of a Low-Fat Meal and Multiple Doses of Ciprofloxacin on the Pharmacokinetics of Vorasidenib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Servier Bio-Innovation LLC (Industry)
Collaborators: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PKH-95032-009
Record Dates: First submitted 2023-04-19; First posted 2023-05-06 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — vorasidenib; Tablets; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: The substudy A (low-fat meal) is an open-label, randomized, balanced, single-dose, 2-treatment, 2-period, crossover study designed to assess the effect of a low-fat meal on the PK following a single oral dose of 40 mg vorasidenib in healthy adult subjects.
  The substudy B (CYP1A2 inhibition) is an open-label, nonrandomized, 2-period, 1-sequence crossover study designed to evaluate the effect of multiple-dose ciprofloxacin (strong CYP1A2 inhibitor) on the single-dose PK of vorasidenib in 28 healthy adult subjects
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Fasting condition / Low-fat meal (Experimental): A single oral dose of 1×40 mg vorasidenib tablet administered under fasted conditions or following a low-fat meal.
  Interventions: Drug: Vorasidenib 40 mg Oral Tablet
- Low-fat meal / Fasted condition (Experimental): A single oral dose of 1×40 mg vorasidenib tablet administered following a low-fat meal or under fasted conditions.
  Interventions: Drug: Vorasidenib 40 mg Oral Tablet
- Vorasidenib (Experimental): Single oral dose of vorasidenib 2×10 mg tablets administered on Day 1.
  Interventions: Drug: Vorasidenib 10 mg Oral Tablet
- Vorasidenib and ciprofloxacin (Experimental): Single oral dose of vorasidenib 2×10 mg tablets administered on Day 1 and twice daily (morning and evening) oral doses of ciprofloxacin 1×500 mg tablet on Days 1 through 14.
  Interventions: Drug: Ciprofloxacin 500 mg Oral Tablet; Drug: Vorasidenib 10 mg Oral Tablet

INTERVENTIONS:
Drug: Vorasidenib 40 mg Oral Tablet — Single oral dose of 1×40 mg vorasidenib tablet administered :
  * under fasted conditions (all subjects will fast overnight for at least 10 hours prior to dosing and for at least 4 hours after dosing.
  * or following a low fat meal (approximatively 400 to 500 calories) (Substudy A)
  Arms: Fasting condition / Low-fat meal; Low-fat meal / Fasted condition
Drug: Ciprofloxacin 500 mg Oral Tablet — Twice daily (morning and evening) oral doses of ciprofloxacin 1×500 mg tablet on Days 1 through 14 (Substudy B)
  Arms: Vorasidenib and ciprofloxacin
Drug: Vorasidenib 10 mg Oral Tablet — Single oral dose of vorasidenib 2×10 mg tablets administered on Day 1 (Substudy B)
  Arms: Vorasidenib; Vorasidenib and ciprofloxacin

SUMMARY:
The objectives of this study are:

* To evaluate the effect of a low-fat meal on the pharmacokinetics (PK) of vorasidenib following a single oral dose of 40 mg vorasidenib in healthy adult subjects (substudy A)
* To evaluate the effect of multiple-dose ciprofloxacin (strong cytochrome P450 [CYP]1A2 inhibitor) on the single-dose PK of vorasidenib in healthy adult subjects (substudy B)

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or non-pregnant, non-lactating female 18 to 55 years of age, inclusive.
2. The subject has a body mass index 18 to 32 kg/m2, inclusive, at screening.
3. The subject has normal hepatic function (aspartate transaminase [AST], alanine transaminase [ALT], total and direct bilirubin, international normalized ratio [INR] all ≤ upper limit of normal [ULN]).
4. The subject has normal renal function as evidenced by creatinine clearance >90 mL/min based on the Cockcroft-Gault glomerular filtration rate estimation: (140 - Age) × (Weight in kg) × (0.85 if female) / (72 × serum creatinine).
5. The subject is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening and check-in.
6. Female subjects of childbearing potential must use 2 effective methods of birth control (eg, diaphragm with spermicide, intrauterine device, condom with foam or vaginal spermicide) or abstinence [true abstinence when this is in line with the preferred and usual lifestyle of the subject]) during the study and for 90 days after the last dose of vorasidenib or be surgically sterile (eg, hysteroscopic sterilization, bilateral tubal ligation or bilateral salpingectomy, hysterectomy, or bilateral oophorectomy), or postmenopausal (defined as amenorrhea 12 consecutive months and documented plasma follicle-stimulating hormone level >40 IU/mL). Female subjects must have a negative pregnancy test at screening and before the first dose of study drug.
7. Male subjects with female partners of childbearing potential must be sterile or be willing to use 2 effective methods of birth control from screening until at least 90 days after the last dose of study drug, or practice abstinence during the study and for 90 days after the last dose of study drug. Abstinence is acceptable only as true abstinence when this is in line with the preferred and usual lifestyle of the subject. Male subjects should also agree to not donate sperm for the duration of the study and until at least 90 days after the last dose of study drug.
8. The subject is a continuous nonsmoker who has not used nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) for at least 3 months prior to the first dose of study drug, based on cotinine test result.
9. The subject agrees to comply with all protocol requirements for the duration of the study.
10. The subject is able to provide written informed consent prior to any procedure required by the study.

Exclusion Criteria:

1. The subject has a history or clinical manifestations of a significant neurological, renal, cardiovascular, gastrointestinal, hepatic, pulmonary, hematologic, immunologic, or psychiatric disease that would preclude study participation, as judged by the investigator.
2. The subject has a history (within 5 years prior to screening) or presence of malignancy, except for adequately treated basal cell and squamous cell carcinoma of the skin.
3. The subject has a history of severe and/or uncontrolled ventricular arrhythmias, or other factors that increase the risk of QT prolongation or arrhythmic events (eg, heart failure, hypomagnesemia, hypokalemia, family history of long QT interval syndrome) or the subject was taking medications that are known to prolong the QT interval unless they can be safely discontinued ≥30 days or 5 half-lives (whichever is longer) before dosing.
4. The subject has any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, and excretion (eg, cholecystectomy, bariatric procedure). Subjects with appendectomy may be included.
5. The subject is a woman of childbearing potential who is pregnant, lactating, or planning to become pregnant within 90 days after the last dose of study drug, or the subject is on oral contraceptive pills (moderate CYP1A2 inhibitors) within 14 days or 5 half-lives (whichever is longer) prior to the first dose administration and/or during the study.
6. The subject has a positive test result for hepatitis B surface antigen or antibodies to hepatitis C virus (HCV) (if antibody test result is positive, it will be followed up with an HCV RNA test to confirm; those with undetectable HCV RNA will not be excluded).
7. The subject has a positive test result for human immunodeficiency virus (HIV) type 1 or 2 antibodies at screening.
8. The subject has a positive test result for the presence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at check-in (Day -1). The subject has received the coronavirus disease 2019 (COVID-19) vaccine within 7 days prior to screening or plans to receive a COVID-19 vaccine within 7 days after receiving the study drug.
9. The subject has used strong CYP1A2 inhibitors and/or inducers within 14 days or 5 half-lives, whichever is longer, prior to the first dose administration and during the study (with the exception of study-specified ciprofloxacin during the study for subjects on Substudy B).
10. The subject has received any vaccine or used any prescription (including hormonal birth control) or over-the-counter medications (except acetaminophen/paracetamol [up to 2 g per day]), including herbal or nutritional supplements, within 30 days or 5 drug half-lives whichever is longer (for all vaccines/medications other than hormonal birth control), or within 14 days or 5 drug half-lives, whichever is longer (for hormonal birth control medications), before the first dose of study drug and throughout the study. Hormone replacement therapy will not be allowed.
11. The subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange-containing products (eg, marmalade), or caffeine- or xanthine-containing products within 48 hours before the first dose of study drug.
12. The subject has a history of symptomatic hypoglycemia or hypoglycemia requiring intervention.
13. The subject has a history of alcoholism or drug abuse within 3 months before screening, or excessive alcohol consumption (regular alcohol intake >21 units per week for male subjects and >14 units of alcohol per week for female subjects) (1 unit is equal to approximately ½ pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits).
14. The subject has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at screening or before the first dose of study drug.
15. The subject is unable or unwilling to abstain from recreational drugs, alcohol, caffeine, xanthine-containing beverages or food (eg, coffee, tea, chocolate, and caffeinated sodas, colas), grapefruit, grapefruit juice, Seville oranges, or products containing any of these, from 48 hours prior to study drug dosing until EOS.
16. The subject has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
17. The subject is involved in strenuous activity (>30 min per day) or contact sports within 48 to 72 hours before dosing and during the study.
18. The subject has excessive exposure to natural or artificial sunlight (tanning beds or UV A/B treatment) within 48 to 72 hours before dosing and during the study.
19. The subject has donated blood or blood products >450 mL within 30 days before the first dose of study drug.
20. The subject has a history of any hypersensitivity, allergy, or other contraindication to the components of the vorasidenib, ciprofloxacin, or activated charcoal formulations used in this study or any significant food allergy.
21. The subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
22. The subject is part of the clinical staff personnel or a family member of the clinical site staff.
23. In the opinion of the investigator, the subject is not suitable for entry into the study.

    Additional Exclusion Criteria for Substudy B:
24. The subject has hypersensitivity to any fluoroquinolone.
25. The subject is at increased risk of Clostridium difficile (eg, prior history of C. difficile infection, recent use of systemic antibiotics [oral, intramuscular, or intravenous] in the last 6 months, recent abdominal surgery within 3 months prior to check-in, history of inflammatory bowel disease, or as judged by the investigator).
26. The subject has had any medical condition that has required frequent or repeat course of antibiotics within the last 6 months. (eg recurrent urinary tract infection [UTI], strep pharyngitis, otitis media, or as judged by the investigator).
27. The subject has any history of tendon rupture or known vascular abnormality.
28. The subject is unable or unwilling to abstain from dairy products or mineral fortified drinks (eg, milk, yogurt, calcium-fortified orange juice) from 48 hours prior to study drug dosing until discharge.
29. The subject has useD of glyburide, cyclosporine, didanosine, methotrexate, or probenecid within 30 days prior to Day 1 or within 5 half-lives of Day 1, whichever is longer.
30. The subject is at high risk for QT prolongation, including:

    1. Baseline QTcF ≥ 450 msec
    2. Risk factors for Torsade de Pointes, including hypocalcemia, hypokalemia, hypomagnesemia, sudden death of unknown cause in a close family member (ie, biological mother, father, or siblings), a near drowning episode, a family history of long QT syndrome.
31. The subject has any history of clinically significant photosensitivity, including, but not limited to a history of phototoxic and/or photoallergic reactions to medications as determined by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Cmax of Vorasidenib (substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  Maximum observed plasma concentration of vorasidenib in substudy A
Tmax of Vorasidenib (substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  Time to maximum observed plasma concentration of vorasidenib in substudy A
AUC0-t of Vorasidenib (substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  Area under the plasma concentration versus time curve (AUC) from time 0 to the last quantifiable concentration (AUC0-t) of vorasidenib in substudy A
AUC0-inf of Vorasidenib (substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  AUC from time 0 extrapolated to infinity (AUC0-inf) of vorasidenib in substudy A
Cmax of Vorasidenib (substudy B) | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  Maximum observed plasma concentration of vorasidenib in substudy B
Tmax of Vorasidenib (substudy B) | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  Time to maximum observed plasma concentration of vorasidenib in substudy B
AUC0-t of Vorasidenib (substudy B) | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  Area under the plasma concentration versus time curve (AUC) from time 0 to the last quantifiable concentration (AUC0-t) of vorasidenib in substudy B
AUC0-inf of Vorasidenib (substudy B) | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  AUC from time 0 extrapolated to infinity (AUC0-inf) of vorasidenib in substudy B

SECONDARY OUTCOMES:
T1/2 of Vorasidenib (Substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  Half-life f vorasidenib in substudy A
CL/F of Vorasidenib (Substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  Apparent oral clearance of vorasidenib in substudy A
Vz/F of Vorasidenib (Substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  Apparent volume of distribution of vorasidenib in substudy A
Cmax of AGI-69460 (Substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  Maximum observed plasma concentration of AGI-69460 in substudy A
Tmax of AGI-69460 (substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  Time to maximum observed plasma concentration of AGI-69460 (substudy A)
AUC0-t of AGI-69460 (substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  Area under the plasma concentration versus time curve (AUC) from time 0 to the last quantifiable concentration (AUC0-t) of AGI-69460 (substudy A)
AUC0-inf of AGI-69460 (substudy A) | Day 1 before dosing (0 hour) and at multiple time points up to 504 hours post-dose
  AUC from time 0 extrapolated to infinity (AUC0-inf) of AGI-69460 (substudy A)
T1/2 of vorasidenib (substudy B) | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  Half-life of vorasidenib in substudy B
CL/F of vorasidenib (substudy B) | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  Apparent oral clearance of vorasidenib in substudy B
Vz/f | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  Apparent volume of distribution of vorasidenib in substudy B
Cmax of AGI-69460 (substudy B) | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  Maximum observed plasma concentration of AGI-69460 in substudy B
Tmax of AGI-69460 (substudy B) | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  Time to maximum observed plasma concentration of AGI-69460 (substudy B)
AUC0-t of AGI-69460 (substudy B) | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  Area under the plasma concentration versus time curve (AUC) from time 0 to the last quantifiable concentration of AGI-69460 (substudy B)
AUC0-inf of AGI-69460 (substudy B) | Before dosing and at multiple time points up to 504 hours on Day 22 after administration of vorasidenib.
  AUC from time 0 extrapolated to infinity (AUC0-inf) of AGI-69460 (substudy B)
Cmax of ciprofloxacin (substudy B) | Before dosing on Day 18 and on multiple time points up to 12 h after dosing
  Maximum observed plasma concentration of ciprofloxacin in substudy B
Tmax of ciprofloxacin (substudy B) | Before dosing on Day 18 and on multiple time points up to 12 h after dosing
  Tmax of ciprofloxacine (substudy B)
AUC0-t of ciprofloxacin (substudy B) | Before dosing on Day 18 and on multiple time points up to 12 h after dosing
  Area under the plasma concentration versus time curve (AUC) from time 0 to the last quantifiable concentration of ciprofloxacin (substudy B)
AUC0-12 of ciprofloxacin (substudy B) | Before dosing on Day 18 and on multiple time points up to 12 h after dosing
  Area under the plasma concentration versus time curve (AUC) from time 0 to 12h of ciprofloxacin (substudy B)

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  sponsored by Servier with a first patient enrolled as of 1 January 2004 onwards for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed
URL: http://clinicaltrials.servier.com/